CLINICAL TRIAL: NCT02509988
Title: Nutritional Intervention Preconception and During Pregnancy to Maintain Healthy Glucose Metabolism and Offspring Health "(NiPPeR)"
Brief Title: Nutritional Intervention Preconception and During Pregnancy to Maintain Healthy Glucose Metabolism and Offspring Health
Acronym: NiPPeR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: National University Hospital, Singapore (Other); Auckland UniServices Ltd. (Industry); Institute for Human Development and Potential (IHDP), Singapore (Other); National University of Singapore (Other); Nestec Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 13597; 34104 (Other: Auckland UniServices Ltd.); 2015/00205 (Other: National University Hospital Singapore); U1111-1171-8056 (Other: Universal Trial Number)
Record Dates: First submitted 2015-07-16; First posted 2015-07-28 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Hyperglycemia
Keywords: Nutrition; Glucose metabolism; Body composition
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (study nutritional drink) (Experimental): Study nutritional drink comes in the form of a sachet to mix with water & take twice a day (once in the morning and once in the evening).
  The drink will be taken before the participant becomes pregnant (for up to 1 year) and throughout pregnancy.
  Interventions: Dietary Supplement: Study nutritional drink
- Control (standard nutritional drink) (Active Comparator): Standard nutritional drink comes in the form of a sachet to mix with water & take twice a day (once in the morning and once in the evening).
  The drink will be taken before the participant becomes pregnant (for up to 1 year) and throughout pregnancy.
  Interventions: Dietary Supplement: Standard nutritional drink

INTERVENTIONS:
Dietary Supplement: Study nutritional drink — Study nutritional drink containing a mix of micronutrients, probiotics and myo-inositol.
  Arms: Intervention (study nutritional drink)
Dietary Supplement: Standard nutritional drink — Standard nutritional drink containing a mix of micronutrients.
  Arms: Control (standard nutritional drink)

SUMMARY:
The study aims to assess whether a nutritional drink taken before conception and continuing through pregnancy, assists in the maintenance of healthy glucose metabolism in the mother and promotes offspring health.

DETAILED DESCRIPTION:
It is known that maternal insulin resistance and high blood glucose levels in early pregnancy alter the functioning of the placenta in ways that persistently affect the supply of nutrients and fat in the unborn baby. There is an increasing focus on the need to optimise preconception nutrition but as yet, limited preconception interventions that are recognized as promoting health for the mother and her child.

The Investigators will recruit up to 1800 women, aged 18-38 years, who are planning a pregnancy in the United Kingdom, Singapore and New Zealand with the aim of securing 600 or more pregnancies. The participants will be randomly allocated to receive the standard nutritional drink or the study nutritional drink. Women who conceive between one and twelve months after starting the nutritional drink will be followed through pregnancy and studied with their babies for three years after delivery. Various testing will be carried out at relevant time points. Mothers will undergo blood, urine, hair and cheek swab sampling, dual-energy X-ray absorptiometry (DXA) scans along with body measurements and health and lifestyle questionnaires. Infants will undergo hair, cheek swab, urine and stool sampling along with body measurements, measurements of body composition and a DXA scan. Placental, cord and other perinatal tissues/samples will be collected.

The data collected will allow identification of the contributions of nutritional and lifestyle factors, social and economic status, ethnicity, genetics and metabolomics and gut microbes to maintaining healthy glucose metabolism in pregnancy, enhancing fertility, mood and reproductive outcomes in the mother, and promoting healthy growth, body composition and wellbeing in the children.

The effect of the intervention on the primary outcome will be examined in two special interest groups; i) women who are overweight or obese prior to conception & ii) women with documented evidence of dysglycemia prior to conception.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-38 years
* Planning to conceive within 6 months
* Able to provide written, informed consent
* In Singapore: Chinese, Malay and Indian ethnicity or mixed Chinese/Malay/Indian ethnicity

Exclusion Criteria:

* Pregnant or lactating at recruitment
* Assisted fertility, apart from those taking clomiphene or letrozole alone
* Pre-existing diabetes (type 1 or type 2)
* Oral or implanted contraception currently or in the last month, or with an Intrauterine Contraceptive Device (IUCD) in situ
* On metformin or systemic steroids currently or in the last month
* Known serious food allergy
* Not able to give informed consent
* Women on anticonvulsants (who are treated with high dose B vitamins in pregnancy) currently or in the last month
* On treatment for Human Immunodeficiency Virus (HIV), Hepatitis B or C currently or in the last month

The partners of the women (over 16 years of age) will also be invited to participate in the study. After having gained written informed consent, fathers will have blood, urine, hair sampling, cheek swabs and body measurements taken and will complete a health and a lifestyle questionnaire at one of the visits during pregnancy.

The mother will consent for their babies to have body measurements, buccal, hair, stool samples and allergy testing from birth to 3.5 years.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1729 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance during pregnancy | Pregnancy Oral Glucose Tolerance Test (OGTT) measurement at 24 - 32 weeks gestation

SECONDARY OUTCOMES:
Duration of gestation | Up to 43 weeks, derived from estimated date of conception from menstrual and ultrasound scan data and date of delivery
Pregnancy weight gain and body composition | Up to 36 weeks, between date of first pregnancy visit and late gestation
Postpartum weight retention and body composition | Up to 2 years, between date of delivery and 6,12 and 24 months postpartum
Change in body composition before, during and after gestation | Up to 4 years, between preconception, pregnancy and 2 years postpartum
Clinical pregnancy, pregnancy loss and live birth rates, including median time to conception of those who conceive during the treatment period and proportions conceiving within 3 months, 6 months and a year of commencing the NiPPeR drink | Between recruitment and delivery
Gestational diabetes frequency | Pregnancy OGTT measurement at 24 - 32 weeks gestation
Hypertensive disorders of pregnancy (pregnancy-induced hypertension and pre-eclampsia/eclampsia) | Up to 49 weeks, between conception derived from estimated date of conception from menstrual and ultrasound scan data and date of delivery, and up to 6 weeks after delivery
Nausea and vomiting frequency | Up to 36 weeks, between 7 weeks of gestation and delivery
Other antenatal, perinatal and postnatal complications | Up to 49 weeks, between conception from estimated date of conception derived from menstrual and ultrasound scan data, and up to 6 weeks after delivery
Preconception and antenatal maternal wellbeing/mood (Edinburgh Post-natal Depression Scale and State-Trait Anxiety Inventory) | Up to 2 years, between preconception and delivery
Postnatal maternal wellbeing/mood (Edinburgh Post-natal Depression Scale and State-Trait Anxiety Inventory) | Up to 52 weeks, between date of delivery and infant age 1 year
Mode of labour onset and delivery | Delivery
Neonatal complications and admission to neonatal care facilities | Up to 4 weeks post-delivery
Preconception maternal micronutrient status (blood analysis) | Date of second preconception visit up to 1 year before pregnancy
Antenatal maternal micronutrient status (blood analysis) | Up to 30 weeks, between 7 weeks gestation and 37 weeks of gestation
Preconception maternal gut microbiota composition and activity profile (analysis of sequencing and transcription data) | Up to 6 weeks from the start of intervention, date of preconception visit 2 which is up to 1 year before pregnancy
Antenatal and postnatal maternal gut and epithelial microbiota composition profile (analysis of sequencing data) | Up to 18 months, between 7 weeks gestation and post-delivery visits
Maternal preconception biochemical, metabolic and molecular profiles | Up to 6 weeks from the start of intervention, date of second preconception visit which is up to 1 year before pregnancy
Maternal antenatal biochemical, metabolic and molecular profiles | Up to 30 weeks, between 7 weeks gestation and 37 weeks of gestation
Placental and cord tissue, and their cellular derivatives: biochemical, metabolic and molecular profiles | Birth
Maternal postnatal biochemical, metabolic and molecular profiles | 6 months after delivery
Maternal preconception epigenetic profile | Preconception to up to 1 year before pregnancy
Maternal antenatal epigenetic profile | Up to 30 weeks, between 7 weeks gestation and 37 weeks of gestation
Maternal postnatal epigenetic profile | 6 months after delivery
Breast milk macronutrient profile (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
Breast milk micronutrient profile (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
Breast milk immune factor profile (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
Breast milk epigenetic profile (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
Breast milk biochemical, metabolic, microbiome and molecular profiles (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
Healthy lactogenesis | Up to 1 year, between date of delivery and 1 year postpartum
Maternal and infant transcriptomics (including of breastmilk) | Up to 34 months, between preconception, pregnancy and 1 year postpartum
Intrauterine growth and wellbeing as assessed by antenatal serial ultrasound scans | Up to 30 weeks, between 7 weeks gestation and 37 weeks of gestation
Offspring birthweight and size at birth | At birth
Offspring size for gestational age at birth, less than the 10th, 10th - 90th, and above the 90th percentiles for gestational age | At birth
Offspring size for gestational age and sex at birth (percentile and standard deviation scores) | At birth
Offspring adiposity (skinfold thicknesses, regional, total and percentage fat mass) | Up to 3.5 years, between date of delivery and 3.5 years postpartum
Adiposity gain, body composition and linear growth during infancy and childhood | Up to 3.5 years, from birth to infant age 3.5 years
Cord blood C-peptide | At delivery
Offspring cardiometabolic profile | Up to 3.5 years, from birth to infant age 3.5 years
Offspring allergic wellbeing | Up to 3.5 years, from birth to infant age 3.5 years
Offspring biochemical, metabolic and molecular profiles | Up to 3.5 years, from birth to infant age 3.5 years
Offspring epigenetic profile | Up to 3.5 years, from birth to infant age 3.5 years
Infant gut microbiota composition and activity | Up to 3.5 years, from birth to infant age 3.5 years
Influence of parental and offspring genotype, sociodemography, body composition, metabolism, lifestyle and diet on the above primary and secondary outcomes at baseline and with the intervention | Up to 5.5 years, between preconception, pregnancy and 3.5 years postpartum

OTHER OUTCOMES:
Health economics analysis (cost benefit analysis) | Composite analysis between preconception visit which is up to 1 year before pregnancy and infant age 3.5 years, assessed up to 5.5 years
Offspring neurocognitive and behavioural development (behavioural and Ages & Stages questionnaires) | Up to 3.5 years, from birth to infant age 3.5 years
Offspring respiratory development (absence of respiratory symptoms) | Up to 3.5 years, from birth to infant age 3.5 years
Offspring allergic development (clinical evaluation of atopic disorders and skin prick test reaction diameter) | Up to 3.5 years, from birth to infant age 3.5 years
Offspring health and wellbeing (questionnaires) | Up to 3.5 years, from birth to infant age 3.5 years
Maternal health and wellbeing | Up to 4 years, between preconception visit which is up to 1 year before pregnancy and up to 2 years after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Cutfield, BHB MB ChB DCH MD FRACP, Principal Investigator — The University of Auckland; Shiao-Yng Chan, MBBChir (UK), FRCOG (UK), PhD, Principal Investigator — National University Hospital, Singapore; Keith Godfrey, BM PhD FRCP, Principal Investigator — MRC Lifecourse Epidemiology Unit, University of Southampton
Locations (3):
- The University of Auckland, Auckland, New Zealand
- National University Hospital, Singapore, Singapore
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

REFERENCES:
- [Background] Godfrey KM, Cutfield W, Chan SY, Baker PN, Chong YS; NiPPeR Study Group. Nutritional Intervention Preconception and During Pregnancy to Maintain Healthy Glucose Metabolism and Offspring Health ("NiPPeR"): study protocol for a randomised controlled trial. Trials. 2017 Mar 20;18(1):131. doi: 10.1186/s13063-017-1875-x. PMID 28320484
- [Derived] Han SM, Huang F, Derraik JGB, Vickers MH, Devaraj S, Redeuil K, Campos-Gimenez E, Pang WW, Godfrey KM, Chan SY, Thakkar SK, Cutfield WS; NiPPeR Study Group. A nutritional supplement during preconception and pregnancy increases human milk vitamin D but not B-vitamin concentrations. Clin Nutr. 2023 Dec;42(12):2443-2456. doi: 10.1016/j.clnu.2023.09.009. Epub 2023 Oct 5. PMID 38411017
- [Derived] Lyons-Reid J, Derraik JGB, Kenealy T, Albert BB, Ramos Nieves JM, Monnard CR, Titcombe P, Nield H, Barton SJ, El-Heis S, Tham E, Godfrey KM, Chan SY, Cutfield WS; NiPPeR Study Group. Impact of preconception and antenatal supplementation with myo-inositol, probiotics, and micronutrients on offspring BMI and weight gain over the first 2 years. BMC Med. 2024 Jan 30;22(1):39. doi: 10.1186/s12916-024-03246-w. PMID 38287349
- [Derived] Godfrey KM, Titcombe P, El-Heis S, Albert BB, Tham EH, Barton SJ, Kenealy T, Chong MF, Nield H, Chong YS, Chan SY, Cutfield WS; NiPPeR Study Group. Maternal B-vitamin and vitamin D status before, during, and after pregnancy and the influence of supplementation preconception and during pregnancy: Prespecified secondary analysis of the NiPPeR double-blind randomized controlled trial. PLoS Med. 2023 Dec 5;20(12):e1004260. doi: 10.1371/journal.pmed.1004260. eCollection 2023 Dec. PMID 38051700
- [Derived] Han SM, Derraik JGB, Vickers MH, Devaraj S, Huang F, Pang WW, Godfrey KM, Chan SY, Thakkar SK, Cutfield WS; NiPPeR Study Group. A nutritional supplement taken during preconception and pregnancy influences human milk macronutrients in women with overweight/obesity and gestational diabetes mellitus. Front Nutr. 2023 Oct 17;10:1282376. doi: 10.3389/fnut.2023.1282376. eCollection 2023. PMID 37915619
- [Derived] Lyons-Reid J, Derraik JGB, Kenealy T, Albert BB, Nieves JMR, Monnard CR, Titcombe P, Nield H, Barton SJ, El-Heis S, Tham E, Godfrey KM, Chan SY, Cutfield WS. The effect of a preconception and antenatal nutritional supplement on children's BMI and weight gain over the first 2 years of life: findings from the NiPPeR randomised controlled trial. Lancet Glob Health. 2023 Mar;11 Suppl 1:S11-S12. doi: 10.1016/S2214-109X(23)00095-5. PMID 36866469
- [Derived] Chan SY, Barton SJ, Loy SL, Chang HF, Titcombe P, Wong JT, Ebreo M, Ong J, Tan KM, Nield H, El-Heis S, Kenealy T, Chong YS, Baker PN, Cutfield WS, Godfrey KM; NiPPeR Study Group. Time-to-conception and clinical pregnancy rate with a myo-inositol, probiotics, and micronutrient supplement: secondary outcomes of the NiPPeR randomized trial. Fertil Steril. 2023 Jun;119(6):1031-1042. doi: 10.1016/j.fertnstert.2023.01.047. Epub 2023 Feb 6. PMID 36754158
- [Derived] Han SM, Devaraj S, Derraik JGB, Vickers MH, Huang F, Dubascoux S, Godfrey KM, Chan SY, Pang WW, Thakkar SK, Cutfield WS; NiPPeR Study Group. A nutritional supplement containing zinc during preconception and pregnancy increases human milk zinc concentrations. Front Nutr. 2023 Jan 10;9:1034828. doi: 10.3389/fnut.2022.1034828. eCollection 2022. PMID 36704795
- [Derived] Lim SX, Cox V, Rodrigues N, Colega MT, Barton SJ, Childs CE, Conlon CA, Wall CR, Cutfield WS, Chan SY, Godfrey KM, Chong MF; NiPPeR Study Group. Evaluation of Preconception Dietary Patterns in Women Enrolled in a Multisite Study. Curr Dev Nutr. 2022 Jun 25;6(7):nzac106. doi: 10.1093/cdn/nzac106. eCollection 2022 Jul. PMID 36628060
- [Derived] Godfrey KM, Barton SJ, El-Heis S, Kenealy T, Nield H, Baker PN, Chong YS, Cutfield W, Chan SY; NiPPeR Study Group. Myo-Inositol, Probiotics, and Micronutrient Supplementation From Preconception for Glycemia in Pregnancy: NiPPeR International Multicenter Double-Blind Randomized Controlled Trial. Diabetes Care. 2021 May;44(5):1091-1099. doi: 10.2337/dc20-2515. Epub 2021 Mar 29. PMID 33782086
- See also: Study Website — http://www.nipperstudy.com